CLINICAL TRIAL: NCT01408381
Title: Multicenter Phase II, Randomized Open Clinical Trial on the Therapeutic Use of Intra-arterial Infusion of Autologous Bone Marrow Mononuclear Cells in Non-diabetic Patients With Critical Chronic Ischemia of Lower Limbs (CLI).
Brief Title: Intra-arterial Infusion of Autologous Bone Marrow Mononuclear Cells in Non-diabetic Patients With Critical Limb Ischemia (CLI).
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Andalusian Initiative for Advanced Therapies - Fundación Pública Andaluza Progreso y Salud (Other)
Collaborators: Iniciativa Andaluza en Terapias Avanzadas (Other)
Responsible Party: Sponsor
Organization: Andalusian Network for Design and Translation of Advanced Therapies (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CMMo/ICC/2009; 2009-013636-20 (EudraCT Number)
Record Dates: First submitted 2011-08-01; First posted 2011-08-03 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2016-03

CONDITIONS: Critical Limb Ischemia (CLI)
Keywords: Critical Limb Ischemia (CLI); Cell Therapy; Bone marrow mononuclear cells
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Control (No Intervention): No cell therapy
- Low dose (Experimental): Intraarterial Infusion of Autologous Bone Marrow Mononuclear Cells: 1 x 108
  Interventions: Other: Intraarterial Infusion of Autologous Bone Marrow Mononuclear Cells
- Intermediate dose (Experimental): Intraarterial Infusion of Autologous Bone Marrow Mononuclear Cells: 5 x 108
  Interventions: Other: Intraarterial Infusion of Autologous Bone Marrow Mononuclear Cells
- High dose (Experimental): Intraarterial Infusion of Autologous Bone Marrow Mononuclear Cells: 1 x 109
  Interventions: Other: Intraarterial Infusion of Autologous Bone Marrow Mononuclear Cells

INTERVENTIONS:
Other: Intraarterial Infusion of Autologous Bone Marrow Mononuclear Cells — Autologous bone marrow-derived mononuclear cells will be infused by an intraarterial catheter into de ischemic limb. The number of infused cells will be 1x108, 5x108 and 1x109 low, intermediate and high dose in the arms respectively.
  Arms: High dose; Intermediate dose; Low dose

SUMMARY:
Phase II Clinical Trial, a prospective, multicenter, open, randomized, parallel-group controlled with three levels of dose.

The hypothesis of the test we propose is that the mononuclear cells of bone marrow provide progenitor cells with regenerative capacity and besides secrete several angiogenic factors, and their implantation into ischemic tissues with both elements should contribute to angiogenesis and tissue regeneration with recovery of the circulation in the affected limb.

DETAILED DESCRIPTION:
The study population will consist of a total of 44 non-diabetic patients with chronic critical ischemia in at least one of their lower limbs (CLI) and without possibility of revascularization. In the experimental group will be included a total of 33 patients divided into three levels of dose, 11 patients in each level (increasing dose of mononuclear cells from autologous bone marrow) and other 11 patients in control group.

* 11 patients in group 1 will not receive cell therapy, and they will only receive conventional treatment, acting as a control group.
* 11 patients in group 2 will receive 1x108 autologous bone marrow mononuclear cells.
* 11 patients in group 3 will receive 5x108 autologous bone marrow mononuclear cells.
* 11 patients in group 4 will receive 1x109 autologous bone marrow mononuclear cells.

The cell therapy drug will be administered intra-arterially in all cases. Patients will be evaluated by clinical, radiological and angiological methods (ankle / brachial pressure index, transcutaneous oxygen pressure, perimeter calf muscle, presence of ulcers, oximetry and digital arteriography).

Patients will receive concomitant drug treatment established by the good clinical practice, so undoubtedly it could be possible that some improvement occurs due to drug treatment.

It is estimated that the inclusion period is approximately 42 months, and the follow-up of each patient of six months. Therefore the total duration of the study will be about forty eight months from the entry of the first patient to the end of the follow-up period of the last patient included.

The primary variable is the improvement in the vascularisation of the treated limb determined by clinical, angiographic and angiologist parameters.

Study objectives :

• Main objective: To evaluate the safety and feasibility of the autotransplantation of autologous bone marrow mononuclear cells administered intra-arterially in non-diabetic patients with critical chronic ischemia of the lower limbs without possibility of either revascularization or other therapeutic alternatives.

Secondary objectives:

1. To compare the effect of three increasing dose of mononuclear cells from autologous bone marrow in the recovery of clinical, angiographic angiologist parameters in non-diabetic patients with critical chronic ischemia of lower limbs to a control group that will have been applied to a conventional treatment.
2. To analyze complications from regenerative therapy itself, from the route of administration and / or study procedures.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes aged ≥ 18 and ≤ 89 years.
* Non-diabetic.
* Infrapopliteal atherosclerotic vascular disease with severe to severe claudication or Rutherford-Becker grade I-3, II, III, in at least one lower limb. The chronic critical ischemia of the lower limb is defined as persistent / recurring pain requiring analgesia and / or non-healing ulcers present> 4 weeks, with no evidence of improvement with conventional therapies and / or walking test (stress test) between 1-6 minutes two exercise tests separated by at least 2 weeks and / or ankle-brachial index at rest <0.8.
* Inability to endovascular or surgical revascularization as recommended by the TransAtlantic Inter-Society Consensus (TASC).
* Failure of the revascularization surgical performed at least 30 days before, either persistently or entry in critical ischemia phase.
* Life expectancy> 2 years.
* Not expected major amputation in the limb to treat in the next 6 months after inclusion.
* Normal laboratory parameters, defined by:

  1. Leukocytes ≥ 3000
  2. Neutrophils ≥ 1500
  3. Platelets ≥ 100,000
  4. Aspartate aminotransferase AST) / Alanine aminotransferase (ALT) ≤ 2.5 standard range institution.
  5. Creatinine ≤ 2.5 mg / dl
* Patients should give their written informed consent to participate in the study.
* Women of childbearing potential must have negative results on a pregnancy test following standard procedures for each hospital performed at the time of inclusion in the study and agree to use a medically approved method of contraception through the duration of the study.

Exclusion Criteria:

* History of malignancy or hematologic disease (myeloproliferative disease, myelodysplastic syndrome or leukemia)
* Patients with uncontrolled hypertension (defined as blood pressure> 180/110 on more than one occasion).
* Severe heart failure (New York Heart Association IV).
* Patients with malignant ventricular arrhythmias or unstable angina.
* Diagnosis of deep vein thrombosis in the previous 3 months.
* Active infection or gangrene wet day infusion of mononuclear bone marrow cells.
* Corporal mass index (BMI)> 40 kg/m2.
* Patients with a diagnosis of alcoholism at the time of inclusion.
* Proliferative retinopathy.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2011-01; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Adverse events | 6 months

SECONDARY OUTCOMES:
Ankle-brachial index | 1 month, 3 months, 6 months
Transcutaneous oxygen pressure (TcO2) | 1 month, 3 months, 6 months
Greater ulcer size | 1 month, 3 months, 6 months
  Ulcer diameter will be recorded
Degree of Rutherford-Becker | 1 month, 3 months, 6 months
Perimeter calf muscle | 1 month, 3 months, 6 months
Presence of faster opacity in infrapopliteal vessels at 6 months compared with the basal situation of the patient. | 1 month, 3 month, 6 month

CONTACTS AND LOCATIONS:
Overall Officials: Inmaculada Herrera, MD, PhD, Study Chair — University Hospital Reina Sofía, Córdoba.; Antonio Chacon, MD, PhD, Principal Investigator — University Hospital Reina Sofia, Córdoba; Diego Martinez, MD, PhD, Principal Investigator — University Hospital Morales Meseguer, Murcia; Jose P Linares, MD, PhD, Principal Investigator — University Hospital San Cecilio, Granada; Vicente Garcia, MD, PhD, Principal Investigator — University Hospital Virgen de las Nieves, Granada; Andres Garcia, MD, PhD, Principal Investigator — University Hospital Nuestra Señora de Valme, Sevilla; Manuel Piñero, MD, PhD, Principal Investigator — University Hospital Puerta del Mar, Cádiz; Fernando Calleja, MD, PhD, Principal Investigator — University Hospital Carlos Haya, Málaga
Locations (5):
- Spain (5):
  - University Hospital Reina Sofía, Córdoba, Cordoba
  - University Hospital Puerta del Mar, Cadiz, Cádiz
  - University Hospital Virgen de las Nieves, Granada, Granada
  - University Hopistal Carlos Haya, Málaga, Málaga
  - University Hospital Nuestra Señora de Valme, Seville, Sevilla

REFERENCES:
- See also: Andalusian Molecular Biology and Regenerative Medicine Centre — http://www.cabimer.es